CLINICAL TRIAL: NCT01608672
Title: Long-Term Patient Satisfaction of Facial Aesthetic Treatment With BOTOX®
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTXC-11-004
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Botulinum toxin Type A (BOTOX®) treatment to glabellar lines as prescribed by the Investigator over at least 5 years.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A (BOTOX®) treatment to glabellar lines as prescribed by the Investigator over at least 5 years.
  Other Names: BOTOX®; OnabotulinumtoxinA; BOTOX® Cosmetic; Vistabel®

SUMMARY:
This is an observational study assessing patient satisfaction following at least 5 years of BOTOX® treatment for glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* At least one BOTOX® treatment for facial wrinkles (glabellar lines) per calendar year for ≥5 years

Exclusion Criteria:

* Received botulinum toxin formulations other than BOTOX®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated for at least 5 years with BOTOX® for glabellar lines
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (5):
- Coral Gables, Florida, United States
- South Yarra, Australia
- São Paulo, Brazil
- Niagara Falls, Ontario, Canada
- Cannes, France

REFERENCES:
- [Background] Trindade de Almeida A, Carruthers J, Cox SE, Goldman MP, Wheeler S, Gallagher CJ. Patient satisfaction and safety with aesthetic onabotulinumtoxinA after at least 5 years: a retrospective cross-sectional analysis of 4,402 glabellar treatments. Dermatol Surg. 2015 Jan;41 Suppl 1:S19-28. doi: 10.1097/DSS.0000000000000275. PMID 25548841

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible patients were identified by retrospective chart review. Demographic and Outcome Measure data were collected at a study visit on Day 1 (approximately 4-28 weeks following last treatment) for patients who received treatment with BOTOX® for ≥5 years. Adverse Event data was collected by retrospective chart review.
Groups:
- All Participants: Botulinum toxin Type A (BOTOX®) treatment to glabellar lines as prescribed by the Investigator over a period of at least 5 years.
Period: Overall Study
Arm/Group | All Participants
Started | 207
Completed | 207
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Mostly or Very Satisfied With Their Glabellar Lines on the Facial Line Satisfaction Questionnaire (FLSQ)
Description: Participants assessed their overall satisfaction with their glabellar lines by answering FLSQ Question 5: "How satisfied are you with the effect your treatment had on your facial lines?" using a 5-point scale where: -2=very dissatisfied, -1=mostly dissatisfied, 0=neither dissatisfied nor satisfied, 1=mostly satisfied and 2=very satisfied. The percentage of participants mostly or very satisfied is reported.
Time Frame: Study Day 1 (approximately 4-28 weeks following last treatment)
Population: Per Protocol population included all enrolled participants who met eligibility criteria with data available for analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 194
Percentage of participants | 92.3

2. Secondary Outcome: Percentage of Participants Mostly or Very Satisfied With Effectiveness of ≥ 5 Years BOTOX® Treatments Using the Patient Questionnaire
Description: Participants rated their overall satisfaction with BOTOX® treatment by answering the question on the Patient Reported Overall Satisfaction of Effectiveness Questionnaire: "You have received BOTOX® facial aesthetic treatment(s) for at least 5 years. How satisfied overall are you with the effect of BOTOX®?" using the following possible answers: Very Dissatisfied, Mostly Dissatisfied, Neither Satisfied or Dissatisfied, Mostly Satisfied or Very Satisfied. The percentage of participants who answered Mostly Satisfied or Very Satisfied is reported.
Time Frame: Study Day 1 (approximately 4-28 weeks following last treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 194
Percentage of participants | 95.8

3. Secondary Outcome: Percentage of Participants Where Physician Was Mostly or Very Satisfied With Effectiveness of ≥ 5 Years BOTOX® Treatments Using the Physician Questionnaire
Description: Physicians rated their overall satisfaction with BOTOX® treatment by answering the question on the Physician Reported Overall Satisfaction of Effectiveness Questionnaire: "You have treated this patient with BOTOX® facial aesthetic treatment(s) for at least 5 years. How satisfied overall are you with the effect of BOTOX®?" using the following possible answers: Very Dissatisfied, Mostly Dissatisfied, Neither Satisfied or Dissatisfied, Mostly Satisfied or Very Satisfied. The percentage of participants where the physician answered Mostly Satisfied or Very Satisfied is reported.
Time Frame: Study Day 1 (approximately 4-28 weeks following last treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 194
Percentage of participants | 98.0

ADVERSE EVENTS:
Time Frame: The collection period was up to 17 years.
Description: Adverse Event data was collected by retrospective chart review. Only treatment related adverse events were reported.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/207
Other Adverse Events (participants affected / at risk) | 23/207
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=207)
Facial paresis (Nervous system disorders) | 23 — Includes lip and mouth asymmetry and brow ptosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.